CLINICAL TRIAL: NCT04581382
Title: Radiation Therapy, Plasma Exchange, and Immunotherapy in Melanoma
Brief Title: Radiation Therapy, Plasma Exchange, and Immunotherapy (Pembrolizumab or Nivolumab) for the Treatment of Melanoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC200703; NCI-2020-06970 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC200703 (Other: Mayo Clinic); R21CA259236 (NIH); 20-003367 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-09-18; First posted 2020-10-09 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; pembrolizumab; Radiotherapy; Radiation; tetraethylpyrazine; Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (radiation therapy, plasma exchange, immunotherapy) (Experimental): Patients undergo radiation therapy daily on days 1-5 (weekdays). Patients then undergo therapeutic plasma exchange over 1-2 hours on the first session starting on the last day of radiation therapy and the last session ending prior to immunotherapy. Beginning day 5, patients receive pembrolizumab IV or nivolumab IV. Treatment with pembrolizumab continues every 3 weeks or treatment with nivolumab continues every 2 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection throughout the study and SOC CT, PET, and/or MRI scans as clinically indicated during follow-up.
  Interventions: Biological: Nivolumab; Biological: Pembrolizumab; Radiation: Radiation Therapy; Biological: Therapeutic Exchange Plasma; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Biological: Therapeutic Exchange Plasma — Undergo therapeutic plasma exchange
  Other Names: TEP
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT SCAN; tomography
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); positron emission tomography scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRS Scan; MRIs; NMR Imaging; NMRI; nuclear magnetic resonance imaging; sMRI; Structural MRI

SUMMARY:
This early phase I trial investigates how well radiation therapy, plasma exchange, and pembrolizumab or nivolumab work in treating patients with melanoma. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Plasma exchange (also known as "plasmapheresis") is a way to "clean" or "flush out" the blood. Immunotherapy with monoclonal antibodies, such as pembrolizumab and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Plasma exchange may help to improve the effect of standard radiation therapy and immunotherapy treatment on tumor cells of patients with melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the kinetics of soluble (s)PD-L1 removal and regeneration by plasma exchange in patients with melanoma.

SECONDARY OBJECTIVES:

I. To observe response at 3 months after plasma exchange plus immunotherapy. II. To observe ongoing response at approximate 3 month intervals after plasma exchange plus immunotherapy.

CORRELATIVE RESEARCH OBJECTIVES:

I. To determine the effects of plasma exchange on immune cell function. II. To observe the kinetics of extracellular vesicles (EVs) after plasma exchange in patients with melanoma.

OUTLINE:

Patients undergo radiation therapy daily on days 1-5 (weekdays). Patients then undergo therapeutic plasma exchange over 1-2 hours on the first session starting on the last day of radiation therapy and the last session ending prior to immunotherapy. Beginning day 5, patients receive pembrolizumab intravenously (IV) or nivolumab IV. Treatment with pembrolizumab continues every 3 weeks or treatment with nivolumab continues every 2 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection throughout the study and standard of care (SOC) computed tomography (CT), positron emission tomography (PET), and/or magnetic resonance imaging (MRI) scans as clinically indicated during follow-up.

After completion of study treatment, patients are followed up at 3 weeks and then for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of melanoma. Patients may have completed biopsy outside of Mayo Clinic, but there must be an internal review done to confirm diagnosis prior to confirming eligibility
* Measurable or non-measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 3
* sPD-L1 levels > 1.7 ng/ml by enzyme-linked immunosorbent assay (ELISA)
* Negative pregnancy test done =< 7 days prior to radiation therapy, for women of childbearing potential only
* Provide written informed consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)
* Willing to provide blood samples for correlative research purposes

Exclusion Criteria:

* Persons taking a biotin supplement
* sPD-L1 level < 1.7 ng/ml by ELISA
* Pregnant or nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2024-10-06 (Actual); Study Completion 2024-10-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of treatment approach | Up to 2 years
  Feasibility will be assessed by being able to complete the study accrual in a reasonable time period.
Kinetics of soluble (s)PD-L1 removal and regeneration by plasma exchange in patients with melanoma | Up to 2 years
  Graphical methods and descriptive statistics will be used to explore this endpoint. Assessed by the change in the sPD-L1 levels over time across the different timepoints of interest.

SECONDARY OUTCOMES:
Overall response rate | Up to 2 years
  Overall response rate is the proportion of patients with a tumor response (partial response or complete response at least 4 weeks apart).
Progression-free survival (PFS) | Up to 2 years
  PFS is defined as the time from registration to the first of either disease progression or death from any cause.
Overall survival (OS) | Up to 2 years
  OS is defined as the time from registration to death from any cause.
Incidence of adverse events (AEs) | Up to 2 years
  The descriptions and grading scales found in the revised National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting. The maximum grade for each type of AE will be recorded for each patient.

OTHER OUTCOMES:
Effects of plasma exchange on immune cell function | Up to 2 years
Kinetics of extracellular vesicles after plasma exchange in patients with melanoma | Up to 2 years
  Will associate the kinetics with clinical outcome data (response rate, OS, PFS).

CONTACTS AND LOCATIONS:
Overall Officials: Sean S. Park, M.D., Ph.D., Principal Investigator — Mayo Clinic in Rochester; Jacob J. Orme, M.D., Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Davidson TM, Foster N, Lucien F, Markovic S, Dong H, Winters JL, Park SS, Orme JJ. Rescuing Cancer Immunity by Plasma Exchange in Metastatic Melanoma (ReCIPE-M1): protocol for a single-institution, open-label safety trial of plasma exchange to clear sPD-L1 for immunotherapy. BMJ Open. 2022 May 12;12(5):e050112. doi: 10.1136/bmjopen-2021-050112. PMID 35551087
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT04581382/ICF_000.pdf